CLINICAL TRIAL: NCT01653002
Title: Methylation Level of SHOX2 in Endobronchial Ultrasound With Real-time Guided Transbronchial Needle Aspiration for Lung Cancer Staging
Status: Completed | Type: Observational
Sponsor: University Hospital, Essen (Other)
Collaborators: Epigenomics, Inc (Industry)
Responsible Party: Principal Investigator, Kaid Darwiche, Dr. med. Kaid Darwiche, University Hospital, Essen
Other Study IDs: RLK-Epi-1; 11-4921-BO (Other: Ethical Review Board University Clinic Essen)
Record Dates: First submitted 2012-07-23; First posted 2012-07-30 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Lung Cancer With Mediastinal Lymph Node Involvement
Keywords: Lung cancer; EBUS-TBNA; Epigenetics; shox2 protein, human
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lung cancer with lymph node involvement
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
A DNA hypermethylation of the gene locus SHOX2 can be frequently found in lung cancer tissue. The purpose of this study is to determine whether the assessment of the hypermethylation level of SHOX2 in specimens obtained by endosonographic guided bronchoscopy makes a contribution to lung cancer staging.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of lung cancer
* enlarged mediastinal or hilar lymph nodes (>10 mm)

Exclusion Criteria:

* clinical condition which excludes general anesthesia

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with proven or suspcted lung cancer and enlarged mediastinal or hilar lymph nodes
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-02; Primary Completion 2012-02 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Diagnostic Performance of SHOX2 | one Year
  Diagnostic performance of SHOX2 methylation Level as biomarker for lung cancer compared to histologic evaluation of EBUS-TBNA specimen alone.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruhrlandklinik - Universitätsklinikum Essen, Essen, Germany